CLINICAL TRIAL: NCT01166412
Title: CCN009: A Multi-center, Open-label, Randomized, Parallel Group Study to Evaluate the Effects on the Mechanisms of Contraceptive Efficacy and, Secondarily, to Assess the Pharmacokinetic Profile and Safety of Two Progestin-only Patches Containing Different Doses of Levonorgestrel (LNG)
Brief Title: A Multi-center, Open-label, Randomized, Parallel Group Study to Evaluate Pharmacokinetic Profile, Effects on the Mechanisms of Contraceptive Efficacy and Safety of Two Progestin-only Patches Containing Different Doses of Levonorgestrel (LNG)
Acronym: CCN009
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCN009
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Contraception
MeSH Terms: interventions — Body Mass Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose level AG1000-6.5 (Active Comparator)
  Interventions: Drug: levonorgestrel patch with BMI 32 kg/m2 to <40 kg/m2; Drug: levonorgestrel patch with BMI <32 kg/m2
- Dose level AG1000-12.5 (Active Comparator)
  Interventions: Drug: levonorgestrel patch with BMI 32 kg/m2 to <40 kg/m2; Drug: levonorgestrel patch with BMI <32 kg/m2

INTERVENTIONS:
Drug: levonorgestrel patch with BMI 32 kg/m2 to <40 kg/m2 — 6.5mg patch daily for 11 weeks
  Other Names: AG 1000-6.5
  Arms: Dose level AG1000-6.5
Drug: levonorgestrel patch with BMI <32 kg/m2 — 6.5mg patch daily for 11 weeks
  Other Names: AG1000-6.5
  Arms: Dose level AG1000-6.5
Drug: levonorgestrel patch with BMI 32 kg/m2 to <40 kg/m2 — 12.5mg patch daily for 11 weeks
  Other Names: AG1000-12.5
  Arms: Dose level AG1000-12.5
Drug: levonorgestrel patch with BMI <32 kg/m2 — 12.5mg patch daily for 11 weeks
  Other Names: AG1000-12.5
  Arms: Dose level AG1000-12.5

SUMMARY:
WHAT IS THE STUDY PRODUCT? The study product is a contraceptive patch, which has the study drug on the patch. The patch is applied directly to the skin and it contains Levonorgestrel (LNG) in a time-release form. LNG is a hormone that has been tested and been approved by the Food & Drug Administration (FDA) in other forms, for example: contraceptive pills, intrauterine devices (IUDs, which are put in the uterus (womb)) and implants (drug in silicon tubing placed under the skin). The use of LNG in the form of a contraceptive patch makes this an experimental drug because the way the drug will be absorbed in the body is a new technique. This study drug does not contain estrogen and it does not protect against HIV, AIDS, or any other sexually transmitted diseases (STDs).

LNG is a progestin (a type of drug that is like a hormone. Progestins can cause changes at the opening of the uterus (womb), such as thickening of the cervical mucus (fluid). This thickened cervical mucus makes it difficult for the male's sperm to reach and fertilize the woman's egg. Since LNG is being absorbed through your skin from the patch, it is experimental, and it is unknown if this study product will really prevent pregnancy like other progestins.

WHY IS THIS STUDY BEING DONE?

The purpose of this study is to find out:

* How well the patch prevents pregnancy
* How safe the patch is to use every day
* How much study drug needs to be in the patch to make sure that it prevents pregnancy
* How the study drug in the patch affects cervical mucus (fluids)
* How the study drug in the patch affects your rate of ovulation (how often you release an egg)
* How well the patch sticks to your skin, without falling off, for a week at a time
* Whether the patch causes any skin irritation or rash (redness or itchiness)
* Whether the study drug in the patch affects your everyday life and if it causes any side effects.

WHAT DOES THE STUDY INVOLVE? We expect that there will be approximately twenty (20) women at each of the six (6) participating clinics in the study. In total, there will be about 120 women from all over the United States who will be in this study. This study is comparing the effectiveness of two different doses of the study drug (40ug and 75 ug) in the patches. This study is an open-label randomized trial, meaning that you and your study doctor will be aware of the dosage of study drug that you will be given. Randomization means that you will be selected by chance, like tossing a coin or rolling a dice. You have a 50% chance of being in the group that receives the 40ug dose patch or the group that receives 75ug dose patch.

DETAILED DESCRIPTION:
This is a Phase I/II, multi-center, open-label, randomized, parallel group, pharmacokinetic, pharmacodynamic study of the AG1000-6.5 and AG1000-12.5 transdermal contraceptive delivery systems (TCDS) in healthy women followed as an outpatient for up to three 28-day cycles (12 weeks or approximately 3 months). During this study, subjects will receive active treatment with the LNG TCDS patches for 11 weeks, followed by one week of post-treatment assessment. The TCDS is designed for one week of patch wear. This study will be conducted by the National Institute of Child Health and Human Development (NICHD) in its Contraceptive Clinical Trials Network (CCTN) at 6 sites in the USA and will enroll approximately 120 women.

This study will enroll approximately 120 subjects, who will be randomized across all sites into the two treatment groups (~60 subjects at each dose level). The randomization schedule will be further stratified to ensure enrollment of approximately 50% of subjects with BMI >32 kg/m2 and <40 kg/m2 and approximately 50% of subjects with BMI <32 kg/m2 for each dose level.

ELIGIBILITY:
Inclusion Criteria:

* 1. Good general health.
* 2. Aged 18-44 years, inclusive, at the enrollment visit.
* 3. Intact uterus with at least one ovary.
* 4. Pap test within the last 12 months or undergo a Pap test at screening prior to enrollment. If a potential subject states that she has had a Pap test within the last 12 months, then she will need to provide documentation of acceptable test results.
* 5. Cervical mucus score of >7, which is based on the modified Insler scoring system during the screening cycle. The cervical mucus is collected by aspiration and the assessment is based on the modified Insler scoring system (the volume and pH of the mucus are not included in the total scoring) yielding a total possible score of 12 (3, 4).
* 6. Regular menstrual cycles that occur every 28 ± 7 days.

  1. If subject is postpartum or post-abortal (with abortion in second trimester), she will be required to have two normal menstrual cycles prior to screening.
  2. If subject had an abortion in the first trimester, she will be required to have at least one menstrual cycle (two menses) prior to screening.
* 7. Heterosexually abstinent or, if heterosexually active, must have undergone previous tubal sterilization, be in monogamous relationship with a vasectomized partner, or only use male or female condoms (use of condoms that are pre-lubricated with or without spermicide is acceptable) for the entire duration of the study. Use of a spermicide applied separately is not allowed. Cervical caps or diaphragms are not allowed during study participation.
* 8. In the opinion of the investigator, able to comply with the protocol, willing to record requested information in the daily diary, and live within the study site catchment area or within a reasonable distance from the site.
* 9. Understand and sign an IRB approved informed consent form prior to screening activities (including fasting blood draw).
* 10. Willing to refrain from use of skin lotions/creams/gels on area of patch application and not use any vaginal creams, lubricants, gels, or spermicides for 3 days prior to study admission through to the end of the study.
* 11. Agree not to participate in any other clinical trials during the course of this study.

Exclusion Criteria:

Contraindications for enrollment will be the same as those for use of combined hormonal contraceptives as referenced in the World Health Organization (WHO) Medical Eligibility Criteria(MEC category 1 or 2) (1), in addition to contra-indications specific to this clinical trial including:

* 1. Known hypersensitivity or contraindication to progestins.
* 2. Known or suspected pregnancy.
* 3. Prior hysterectomy or bilateral oophorectomy.
* 4. Prior cervical surgery (LEEP, Cone biopsy, Cryosurgery).
* 5. A history (within prior 12 months) or drug or alcohol abuse.
* 6. Undiagnosed abnormal genital bleeding.
* 7. Undiagnosed vaginal discharge or vaginal lesions or abnormalities. Subjects diagnosed at screening with a Chlamydia or gonococcus infection may not be included in the trial unless they are treated and proof of cure is documented after treatment (i.e. repeat test with negative results). In accordance with PI/medical designee assessment and local standards of practice, women with a history of genital herpes can be included if outbreaks are infrequent. Antiviral prophylactic therapy is permitted.
* 8. Uncontrolled thyroid disorder.
* 9. History or presence of dermal hypersensitivity in response to topical application. Specifically any reaction to application of a plastic bandage (Band-Aid), surgical or bandage tape, other skin patches, or adhesives.
* 10. Any Pap test finding that would require additional workup or treatment during the study interval. HPV testing will not be done at screening for these subjects.
* 11. Use of an injectable hormonal contraceptive (Depo-Provera®) within the past 10 months.
* 12. Use of oral contraceptives, contraceptive implants, or other sex steroid hormones within 30 days prior to screening visit.
* 13. Women who are breastfeeding or within 30 days of discontinuing breast feeding.
* 14. Women planning to undergo major surgery within four months of study enrollment.
* 15. Women planning pregnancy within their months of study enrollment.
* 16. Smoking in women who are ages 18-44 years old that smoke 15 cigarettes or more per day must be evaluated by the PI for inclusion based on risk factors that would increase their risk for CVD and thromboembolism.
* 17. Current or past deep vein thrombophlebitis or thromboembolic disorders.
* 18. History of known thrombophilia in a first-degree relative <45 years of age suggesting familial defect in blood coagulation system, which in the opinion of the principal investigator, suggests use of a hormonal contraceptive could pose a significant risk.
* 19. Cerebrovascular or cardiovascular disease or increased risk for arterial thrombosis.
* 20. History of retinal vascular lesions, unexplained partial or complete loss of vision.
* 21. Known or suspected carcinoma of the breast, endometrium, or any other known or suspected progestin-dependent neoplasia.
* 22. Past history of any other carcinoma (excluding basal cell carcinomas) unless in remission for more than 5 years.
* 23. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive, unless she is stable on antidepressant medication.
* 24. Headaches with focal neurological symptoms only in women over 35 years old.
* 25. History of cholestatic jaundice of pregnancy or jaundice with prior steroid use or other benign or malignant liver tumors; active liver disease.
* 26. Systolic BP > 140 mm Hg and/or Diastolic blood pressure (BP) > 90 mm Hg after 5-10 minutes rest.
* 27. Clinically significant abnormal serum chemistry values according to the Principal Investigator's judgment.
* 28. Participation in another clinical trial involving an investigational drug or device within last 30 days (prior to screening).
* 29. Use of liver enzyme inducers within last 90 days (prior to screening) or intention to use liver enzyme inducers during the study (see Appendix 2 Exclusionary Medication List).
* 30. Known HIV infection.
* 31. Women at high risk of contracting HIV, e.g. women with multiple sex partners who need to use condoms consistently, injection drug users. Women enrolled in the study, who use condoms to protect against STIs or pregnancy, should be instructed that they can use condoms that are pre-lubricated with spermicide or lubricated, but they cannot use a spermicide applied separately and they should record all condom use in their diaries.
* 32. Women who use any medications on the Exclusionary Medication List (see Appendix 2) OR used any within the past three months prior to the screening visit.
* 33. Women with BMI ≥40 kg/m2 are excluded.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Colorado - Adv. Repro. Med., Aurora, Colorado
  - Columbia University, New York, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level AG1000-6.5: levonorgestrel patch with BMI <32 kg/m2: 6.5mg patch daily for 11 weeks
  levonorgestrel patch with BMI 32 kg/m2 - <40 kg/m2: 6.5mg patch daily for 11 weeks
- Dose Level AG1000-12.5: levonorgestrel patch with BMI <32 kg/m2: 12.5mg patch daily for 11 weeks
  levonorgestrel patch with BMI 32 kg/m2 - <40 kg/m2: 12.5mg patch daily for 11 weeks
Period: Overall Study
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Started | 61 | 60
Completed | 56 | 48
Not Completed | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5 | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 60 | 121
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (5.92) | 31.0 (7.22) | 30.9 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Poor Cervical Mucus Scores During Treatment Period
Description: The primary endpoint is a subject's incidence of the "Poor" cervical mucus score as determined by the modified Insler score. The cervical mucus score will be based on the modified Insler scoring system (the volume and pH of the mucus are not included in the total scoring) yielding a total possible modified Insler cervical mucus score of 12 (3, 4). The total modified Insler cervical mucus scores of 0-4, 5-8 and 9-12 will be categorized as "Poor," "Fair" and "Good," respectively.
Time Frame: Visit 1 (Treatment Day 1) through Visit 19 (Treatment Day 79)
Population: Only cervical mucus data collected after the first dose of study drug is included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
Participants | 3 | 11

2. Secondary Outcome: Changes From Baseline in Endometrial Thickness
Description: Changes from Baseline in endometrial thickness measured at Visit 1, Visits 3-5, Visits 7-10, Visit 12-18 (Days 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78)
Time Frame: Days 0, 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, up to 78 days
Population: Subjects that had endometrial thickness measured at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
mm
  Baseline | 7.68 (3.243) | 7.90 (2.792)
  Change from Baseline to Visit 1/Day 1 | -2.94 (3.885) | -3.32 (3.730)
  Change from Baseline to Visit 3/Day 5: number analyzed (Participants) | 59 | 55
  Change from Baseline to Visit 3/Day 5 | -2.77 (3.377) | -3.15 (2.936)
  Change from Baseline to Visit 4/Day 8: number analyzed (Participants) | 58 | 57
  Change from Baseline to Visit 4/Day 8 | -1.75 (3.706) | -2.00 (3.121)
  Change from Baseline to Visit 5/Day 11: number analyzed (Participants) | 57 | 57
  Change from Baseline to Visit 5/Day 11 | -0.71 (3.239) | -2.50 (3.673)
  Change from Baseline to Visit 7/Day 18: number analyzed (Participants) | 59 | 56
  Change from Baseline to Visit 7/Day 18 | -0.91 (4.367) | -2.16 (3.216)
  Change from Baseline to Visit 8/Day 22: number analyzed (Participants) | 59 | 55
  Change from Baseline to Visit 8/Day 22 | -1.34 (3.960) | -2.69 (3.384)
  Change from Baseline to Visit 9/Day 25: number analyzed (Participants) | 59 | 53
  Change from Baseline to Visit 9/Day 25 | -1.97 (3.834) | -2.87 (3.769)
  Change from Baseline to Visit 10/Day 29: number analyzed (Participants) | 59 | 54
  Change from Baseline to Visit 10/Day 29 | -2.67 (3.234) | -3.26 (3.413)
  Change from Baseline to Visit 12/Day 36: number analyzed (Participants) | 59 | 53
  Change from Baseline to Visit 12/Day 36 | -2.10 (3.995) | -3.16 (3.436)
  Change from Baseline to Visit 13/Day 43: number analyzed (Participants) | 57 | 52
  Change from Baseline to Visit 13/Day 43 | -1.67 (3.837) | -3.18 (3.183)
  Change from Baseline to Visit 14/Day 50: number analyzed (Participants) | 57 | 49
  Change from Baseline to Visit 14/Day 50 | -1.72 (4.422) | -3.24 (3.456)
  Change from Baseline to Visit 15/Day 57: number analyzed (Participants) | 57 | 49
  Change from Baseline to Visit 15/Day 57 | -2.18 (3.940) | -3.80 (3.477)
  Change from Baseline to Visit 16/Day 64: number analyzed (Participants) | 57 | 47
  Change from Baseline to Visit 16/Day 64 | -2.26 (3.676) | -3.39 (3.637)
  Change from Baseline to Visit 17/Day 71: number analyzed (Participants) | 57 | 49
  Change from Baseline to Visit 17/Day 71 | -2.08 (4.175) | -3.56 (3.224)
  Change from Baseline to Visit 18/Day 78: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 18/Day 78 | -1.95 (3.857) | -2.84 (3.526)

3. Secondary Outcome: Patch Wearability Based on Patch Adhesion
Description: Patch wearability measured by patch adhesion at Visit 4, Visit 6, Visit 8, Visit 10, Visits 12-18 (Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78) based on the following criteria: > 90% = > 90% of patch adhered (no lift from skin); >75% but < 90% = > 75% adhered but < 90% (some edges showing lift from skin); > 50% but < 75% = > 50% adhered but < 75% (half of patch lifts of skin; < 50% = < 50% adherence ( > half of patch lifts off, but not detached); Patch Off = patch completely detached from skin
Time Frame: Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, up to 78 days
Population: subjects that had patch adhesion assessed during the respective timepoints are included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 61 | 60
Participants
  Visit 4/Day 8: >90%: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: >90% | 49 | 50
  Visit 4/Day 8: 75-90%: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: 75-90% | 9 | 7
  Visit 4/Day 8: 50-75%: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: 50-75% | 1 | 0
  Visit 4/Day 8: <50%: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: <50% | 0 | 0
  Visit 4/Day 8: Patch Off: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: Patch Off | 1 | 1
  Visit 6/Day 15: >90%: number analyzed (Participants) | 58 | 57
  Visit 6/Day 15: >90% | 52 | 46
  Visit 6/Day 15: 75-90%: number analyzed (Participants) | 58 | 57
  Visit 6/Day 15: 75-90% | 6 | 9
  Visit 6/Day 15: 50-75%: number analyzed (Participants) | 58 | 57
  Visit 6/Day 15: 50-75% | 0 | 1
  Visit 6/Day 15: <50%: number analyzed (Participants) | 58 | 57
  Visit 6/Day 15: <50% | 0 | 0
  Visit 6/Day 15: Patch Off: number analyzed (Participants) | 58 | 57
  Visit 6/Day 15: Patch Off | 0 | 1
  Visit 8/Day 22: >90%: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: >90% | 54 | 46
  Visit 8/Day 22: 75-90%: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: 75-90% | 4 | 7
  Visit 8/Day 22: 50-75%: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: 50-75% | 0 | 0
  Visit 8/Day 22: <50%: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: <50% | 0 | 1
  Visit 8/Day 22: Patch Off: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: Patch Off | 1 | 1
  Visit 10/Day 29: >90%: number analyzed (Participants) | 58 | 53
  Visit 10/Day 29: >90% | 56 | 44
  Visit 10/Day 29: 75-90%: number analyzed (Participants) | 58 | 53
  Visit 10/Day 29: 75-90% | 2 | 8
  Visit 10/Day 29: 50-75%: number analyzed (Participants) | 58 | 53
  Visit 10/Day 29: 50-75% | 0 | 1
  Visit 10/Day 29: <50%: number analyzed (Participants) | 58 | 53
  Visit 10/Day 29: <50% | 0 | 0
  Visit 10/Day 29: Patch Off: number analyzed (Participants) | 58 | 53
  Visit 10/Day 29: Patch Off | 0 | 0
  Visit 12/Day 36: >90%: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: >90% | 53 | 47
  Visit 12/Day 36: 75-90%: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: 75-90% | 4 | 3
  Visit 12/Day 36: 50-75%: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: 50-75% | 0 | 3
  Visit 12/Day 36: <50%: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: <50% | 0 | 0
  Visit 12/Day 36: Patch Off: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: Patch Off | 2 | 1
  Visit 13/Day 43: >90%: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: >90% | 51 | 46
  Visit 13/Day 43: 75-90%: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: 75-90% | 6 | 4
  Visit 13/Day 43: 50-75%: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: 50-75% | 0 | 1
  Visit 13/Day 43: <50%: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: <50% | 0 | 0
  Visit 13/Day 43: Patch Off: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: Patch Off | 0 | 0
  Visit 14/Day 50: >90%: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: >90% | 55 | 42
  Visit 14/Day 50: 75-90%: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: 75-90% | 2 | 8
  Visit 14/Day 50: 50-75%: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: 50-75% | 0 | 0
  Visit 14/Day 50: <50%: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: <50% | 0 | 0
  Visit 14/Day 50: Patch Off: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: Patch Off | 0 | 0
  Visit 15/Day 57: >90%: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: >90% | 51 | 44
  Visit 15/Day 57: 75-90%: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: 75-90% | 5 | 4
  Visit 15/Day 57: 50-75%: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: 50-75% | 0 | 0
  Visit 15/Day 57: <50%: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: <50% | 0 | 0
  Visit 15/Day 57: Patch Off: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: Patch Off | 1 | 1
  Visit 16/Day 64: >90%: number analyzed (Participants) | 56 | 48
  Visit 16/Day 64: >90% | 51 | 43
  Visit 16/Day 64: 75-90%: number analyzed (Participants) | 56 | 48
  Visit 16/Day 64: 75-90% | 5 | 4
  Visit 16/Day 64: 50-75%: number analyzed (Participants) | 56 | 48
  Visit 16/Day 64: 50-75% | 0 | 0
  Visit 16/Day 64: <50%: number analyzed (Participants) | 56 | 48
  Visit 16/Day 64: <50% | 0 | 0
  Visit 16/Day 64: Patch Off: number analyzed (Participants) | 56 | 48
  Visit 16/Day 64: Patch Off | 0 | 1
  Visit 17/Day 71: >90%: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: >90% | 54 | 45
  Visit 17/Day 71: 75-90%: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: 75-90% | 3 | 4
  Visit 17/Day 71: 50-75%: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: 50-75% | 0 | 0
  Visit 17/Day 71: <50%: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: <50% | 0 | 0
  Visit 17/Day 71: Patch Off: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: Patch Off | 0 | 0
  Visit 18/Day 78: >90%: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: >90% | 53 | 40
  Visit 18/Day 78: 75-90%: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: 75-90% | 3 | 5
  Visit 18/Day 78: 50-75%: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: 50-75% | 0 | 0
  Visit 18/Day 78: <50%: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: <50% | 0 | 0
  Visit 18/Day 78: Patch Off: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: Patch Off | 0 | 3

4. Secondary Outcome: LNG PK Profiles After the First and Fifth Patches Are Applied and After the Eleventh (Last) Patch is Removed
Description: LNG PK at 0, 1, 2, 4, and 6 hours with patch on Day 1 (Visit 1), Day 29 (Visit 5), and Day 78 (Visit 12) after patch removal using Area Under the Curve Mean at each visit. The mean area under the curve represents the amount of LNG in the body at the given timepoint.
Time Frame: Day 1 (Visit 1), Day 29 (Visit 5), and Day 78 (Visit 12), up to 78 days
Population: subjects that had samples collected at the respective timeframes were analyzed
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 61 | 60
hr*pg/mL
  Day 1/Visit 1: number analyzed (Participants) | 60 | 60
  Day 1/Visit 1 | 322.6247 (141.24822) | 401.3429 (200.31346)
  Day 29/Visit 5: number analyzed (Participants) | 54 | 48
  Day 29/Visit 5 | 1326.6995 (1663.88816) | 1997.9708 (1626.87132)
  Day 78/Visit 12 | 945.0963 (590.16226) | 1303.4188 (781.29795)

5. Secondary Outcome: Single Serum LNG PK Measures at Various Times On-treatment and Post Treatment.
Description: Serum LNG measures at Day 2 (Visit 2), Day 8 (Visit 4), Day 15 (Visit 6), Day 22 (Visit 8), Days 30, 36, 43, 50, 57, 64, 71 (Visits 11-17), Days 79, 80, 81, 82, 85 (Visits 19-23)
Time Frame: Treatment Days 2, 8, 15, 22, 30, 36, 43, 50, 57, 64, 71, 79, 80, 81, 82, and 85, up to 85 days
Population: subjects that had samples collected during the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 61 | 60
ng/mL
  Day 2: number analyzed (Participants) | 60 | 57
  Day 2 | 181.489 (174.4023) | 392.703 (354.6305)
  Day 8: number analyzed (Participants) | 59 | 58
  Day 8 | 183.140 (143.5979) | 301.107 (181.3892)
  Day 15: number analyzed (Participants) | 58 | 56
  Day 15 | 175.092 (123.0980) | 290.184 (212.5369)
  Day 22: number analyzed (Participants) | 59 | 55
  Day 22 | 174.769 (126.9624) | 349.906 (259.7689)
  Day 30: number analyzed (Participants) | 57 | 51
  Day 30 | 276.579 (247.4270) | 519.327 (398.7602)
  Day 36: number analyzed (Participants) | 59 | 55
  Day 36 | 178.315 (135.2644) | 309.459 (320.7415)
  Day 43: number analyzed (Participants) | 57 | 53
  Day 43 | 168.591 (136.0588) | 301.725 (218.2762)
  Day 50: number analyzed (Participants) | 57 | 50
  Day 50 | 174.454 (143.7253) | 330.625 (282.0871)
  Day 57: number analyzed (Participants) | 56 | 50
  Day 57 | 176.129 (133.7951) | 272.921 (171.9373)
  Day 64: number analyzed (Participants) | 57 | 47
  Day 64 | 162.538 (130.8442) | 276.387 (198.0998)
  Day 71: number analyzed (Participants) | 56 | 48
  Day 71 | 167.253 (128.7246) | 280.677 (177.6261)
  Day 79: number analyzed (Participants) | 55 | 44
  Day 79 | 100.182 (54.7594) | 129.584 (76.1130)
  Day 80: number analyzed (Participants) | 55 | 45
  Day 80 | 72.311 (41.8869) | 87.295 (53.3175)
  Day 81: number analyzed (Participants) | 55 | 44
  Day 81 | 48.481 (22.9973) | 66.773 (37.6578)
  Day 82: number analyzed (Participants) | 48 | 42
  Day 82 | 37.506 (22.2807) | 49.627 (25.1602)
  Day 85: number analyzed (Participants) | 55 | 45
  Day 85 | 29.554 (25.5765) | 38.882 (38.1462)

6. Secondary Outcome: Changes From Baseline in Estradiol Levels
Description: Changes from Baseline (Visit 1) in Estradiol levels measured at Visits 3-10, Visit 12-18, Visit 23 (Days 0, 5, 8, 11, 15, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, 85)
Time Frame: Days 0, 5, 8, 11, 15, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, 85, up to 85 days
Population: subjects that had samples collected at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
pg/mL
  Baseline | 44.1 (16.61) | 47.2 (48.40)
  Change from Baseline to Visit 3/Day 5: number analyzed (Participants) | 59 | 53
  Change from Baseline to Visit 3/Day 5 | 44.7 (66.19) | 43.8 (60.55)
  Change from Baseline to Visit 4/Day 8: number analyzed (Participants) | 59 | 57
  Change from Baseline to Visit 4/Day 8 | 119.4 (108.95) | 103.2 (138.77)
  Change from Baseline to Visit 5/Day 11: number analyzed (Participants) | 58 | 55
  Change from Baseline to Visit 5/Day 11 | 158.4 (166.04) | 170.7 (207.28)
  Change from Baseline to Visit 6/Day 15: number analyzed (Participants) | 58 | 55
  Change from Baseline to Visit 6/Day 15 | 147.1 (143.95) | 191.9 (249.75)
  Change from Baseline to Visit 7/Day 18: number analyzed (Participants) | 58 | 56
  Change from Baseline to Visit 7/Day 18 | 129.1 (122.25) | 123.8 (164.50)
  Change from Baseline to Visit 8/Day 22: number analyzed (Participants) | 59 | 55
  Change from Baseline to Visit 8/Day 22 | 71.5 (107.17) | 76.6 (120.61)
  Change from Baseline to Visit 9/Day 25: number analyzed (Participants) | 58 | 54
  Change from Baseline to Visit 9/Day 25 | 33.8 (78.86) | 65.0 (121.64)
  Change from Baseline to Visit 10/Day 29: number analyzed (Participants) | 59 | 54
  Change from Baseline to Visit 10/Day 29 | 21.4 (55.67) | 37.8 (98.50)
  Change from Baseline to Visit 12/Day 36: number analyzed (Participants) | 59 | 55
  Change from Baseline to Visit 12/Day 36 | 101.6 (150.53) | 53.9 (110.20)
  Change from Baseline to Visit 13/Day 43: number analyzed (Participants) | 57 | 53
  Change from Baseline to Visit 13/Day 43 | 113.4 (173.71) | 98.6 (172.48)
  Change from Baseline to Visit 14/Day 50: number analyzed (Participants) | 57 | 49
  Change from Baseline to Visit 14/Day 50 | 85.7 (118.49) | 73.7 (166.09)
  Change from Baseline to Visit 15/Day 57: number analyzed (Participants) | 56 | 50
  Change from Baseline to Visit 15/Day 57 | 76.4 (135.90) | 40.1 (117.25)
  Change from Baseline to Visit 16/Day 64: number analyzed (Participants) | 57 | 47
  Change from Baseline to Visit 16/Day 64 | 94.5 (165.60) | 42.4 (104.84)
  Change from Baseline to Visit 17/Day 71: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 17/Day 71 | 82.6 (114.90) | 51.3 (99.92)
  Change from Baseline to Visit 18/Day 78: number analyzed (Participants) | 57 | 48
  Change from Baseline to Visit 18/Day 78 | 73.2 (101.43) | 76.1 (118.96)
  Change from Baseline to Visit 23/Day 85: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 23/Day 85 | 77.1 (119.08) | 78.0 (104.52)

7. Secondary Outcome: Changes From Baseline in Luteinizing Hormone Levels
Description: Changes from Baseline (Visit 1) in LH levels measured at Visits 3-10, Visit 12-18, Visit 23 (Days 0, 5, 8, 11, 15, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, 85)
Time Frame: Days 0, 5, 8, 11, 15, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, 85, up to 85 days
Population: subjects that had samples collected at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
mIU/mL
  Baseline | 4.988 (1.8540) | 5.272 (2.0365)
  Change from Baseline to Visit 3/Day 5: number analyzed (Participants) | 59 | 53
  Change from Baseline to Visit 3/Day 5 | 2.318 (3.1376) | 2.391 (2.3369)
  Change from Baseline to Visit 4/Day 8: number analyzed (Participants) | 59 | 57
  Change from Baseline to Visit 4/Day 8 | 3.647 (3.9407) | 2.855 (3.5869)
  Change from Baseline to Visit 5/Day 11: number analyzed (Participants) | 58 | 55
  Change from Baseline to Visit 5/Day 11 | 5.306 (4.5544) | 3.573 (3.3224)
  Change from Baseline to Visit 6/Day 15: number analyzed (Participants) | 58 | 55
  Change from Baseline to Visit 6/Day 15 | 4.011 (15.0705) | 1.759 (3.4399)
  Change from Baseline to Visit 7/Day 18: number analyzed (Participants) | 58 | 56
  Change from Baseline to Visit 7/Day 18 | 0.193 (4.0425) | -0.024 (4.3170)
  Change from Baseline to Visit 8/Day 22: number analyzed (Participants) | 59 | 55
  Change from Baseline to Visit 8/Day 22 | -0.625 (2.6920) | -0.108 (4.0482)
  Change from Baseline to Visit 9/Day 25: number analyzed (Participants) | 58 | 54
  Change from Baseline to Visit 9/Day 25 | -0.233 (2.5591) | 0.094 (3.6229)
  Change from Baseline to Visit 10/Day 29: number analyzed (Participants) | 59 | 54
  Change from Baseline to Visit 10/Day 29 | 0.071 (1.8310) | 0.597 (3.8260)
  Change from Baseline to Visit 12/Day 36: number analyzed (Participants) | 59 | 55
  Change from Baseline to Visit 12/Day 36 | 2.219 (4.3152) | 1.377 (3.3823)
  Change from Baseline to Visit 13/Day 43: number analyzed (Participants) | 57 | 53
  Change from Baseline to Visit 13/Day 43 | 1.143 (3.1123) | 1.915 (6.8802)
  Change from Baseline to Visit 14/Day 50: number analyzed (Participants) | 57 | 49
  Change from Baseline to Visit 14/Day 50 | -0.146 (2.6963) | 0.918 (3.5897)
  Change from Baseline to Visit 15/Day 57: number analyzed (Participants) | 56 | 50
  Change from Baseline to Visit 15/Day 57 | 0.738 (3.6271) | 0.916 (3.7356)
  Change from Baseline to Visit 16/Day 64: number analyzed (Participants) | 57 | 47
  Change from Baseline to Visit 16/Day 64 | 2.835 (8.3480) | 2.622 (3.8875)
  Change from Baseline to Visit 17/Day 71: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 17/Day 71 | 1.158 (3.3195) | 1.512 (4.0583)
  Change from Baseline to Visit 18/Day 78: number analyzed (Participants) | 57 | 48
  Change from Baseline to Visit 18/Day 78 | 0.302 (4.6718) | 1.335 (4.1741)
  Change from Baseline to Visit 23/Day 85: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 23/Day 85 | 2.780 (8.988) | 1.416 (4.0763)

8. Secondary Outcome: Changes From Baseline in Follicle-Stimulating Hormone Levels
Description: Changes from Baseline (Visit 1) in FSH levels measured at Visits 10/Day 29, Visit 15/Day 57, Visit 18/Day 78, Visit 23/Day 85
Time Frame: Days 0, 29, 57, 78, 85, up to 85 days
Population: subjects that had samples collected at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
mIU/mL
  Baseline: number analyzed (Participants) | 60 | 56
  Baseline | 6.588 (2.1862) | 6.626 (2.5115)
  Change from Baseline to Visit 10/Day 29: number analyzed (Participants) | 60 | 56
  Change from Baseline to Visit 10/Day 29 | -0.928 (1.8646) | -1.368 (2.2185)
  Change from Baseline to Visit 15/Day 57: number analyzed (Participants) | 57 | 50
  Change from Baseline to Visit 15/Day 57 | -1.912 (2.6797) | -1.858 (3.1649)
  Change from Baseline to Visit 18/Day 78: number analyzed (Participants) | 57 | 48
  Change from Baseline to Visit 18/Day 78 | -2.190 (2.6875) | -2.113 (3.0552)
  Change from Baseline to Visit 23/Day 85: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 23/Day 85 | -1.035 (2.4421) | -2.003 (2.8092)

9. Secondary Outcome: Changes From Baseline in Sex Hormone-Binding Globulin Levels
Description: Changes from Baseline (Visit 1) in SHBG levels measured at Visits 10/Day 29, Visit 15/Day 57, Visit 18/Day 78, Visit 23/Day 85
Time Frame: Days 0, 29, 57, 78, 85, up to 85 days
Population: subjects that had samples collected at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
ug/mL
  Baseline: number analyzed (Participants) | 60 | 56
  Baseline | 5.407 (2.5143) | 5.367 (2.3355)
  Change from Baseline to Visit 10/Day 29: number analyzed (Participants) | 59 | 56
  Change from Baseline to Visit 10/Day 29 | -1.243 (1.2113) | -1.737 (1.5096)
  Change from Baseline to Visit 15/Day 57: number analyzed (Participants) | 57 | 50
  Change from Baseline to Visit 15/Day 57 | -1.032 (1.4994) | -2.158 (1.5545)
  Change from Baseline to Visit 18/Day 78: number analyzed (Participants) | 57 | 48
  Change from Baseline to Visit 18/Day 78 | -1.091 (1.3419) | -2.203 (1.5719)
  Change from Baseline to Visit 23/Day 85: number analyzed (Participants) | 56 | 48
  Change from Baseline to Visit 23/Day 85 | -0.585 (1.2964) | -1.299 (1.4768)

10. Secondary Outcome: Ovarian Follicular Activity Measured by the Number of Follicles Greater Than or Equal to 6mm
Description: Number of follicles greater than or equal to 6mm at Baseline, Visits 1-10, Visits 12-18 (Days 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78)
Time Frame: Days 0, 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, up to 78 days
Population: Subjects that had follicles measured and counted were analyzed
Measure: Mean (Standard Deviation); unit: Number of Follicles
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
Number of Follicles
  Baseline: number analyzed (Participants) | 59 | 57
  Baseline | 2.9 (2.59) | 2.9 (2.71)
  Visit 1/Day 1: number analyzed (Participants) | 59 | 57
  Visit 1/Day 1 | 2.5 (2.16) | 2.1 (1.77)
  Visit 3/Day 5: number analyzed (Participants) | 58 | 55
  Visit 3/Day 5 | 3.4 (2.71) | 3.8 (4.64)
  Visit 4/Day 8: number analyzed (Participants) | 57 | 57
  Visit 4/Day 8 | 3.2 (3.05) | 3.1 (3.03)
  Visit 5/Day 11: number analyzed (Participants) | 57 | 57
  Visit 5/Day 11 | 2.7 (1.91) | 2.4 (1.92)
  Visit 7/Day 18: number analyzed (Participants) | 59 | 56
  Visit 7/Day 18 | 1.9 (1.65) | 2.1 (2.05)
  Visit 8/Day 22: number analyzed (Participants) | 58 | 54
  Visit 8/Day 22 | 1.2 (1.31) | 2.4 (4.94)
  Visit 9/Day 25: number analyzed (Participants) | 59 | 53
  Visit 9/Day 25 | 1.6 (1.83) | 2.0 (2.03)
  Visit 10/Day 29: number analyzed (Participants) | 59 | 52
  Visit 10/Day 29 | 2.6 (2.47) | 2.0 (1.58)
  Visit 12/Day 36: number analyzed (Participants) | 59 | 53
  Visit 12/Day 36 | 2.7 (2.84) | 2.6 (2.35)
  Visit 13/Day 43: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43 | 2.4 (2.23) | 2.1 (1.99)
  Visit 14/Day 50: number analyzed (Participants) | 57 | 49
  Visit 14/Day 50 | 1.6 (1.76) | 2.2 (1.71)
  Visit 15/Day 57: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57 | 2.3 (2.14) | 2.9 (3.30)
  Visit 16/Day 64: number analyzed (Participants) | 57 | 47
  Visit 16/Day 64 | 2.6 (2.50) | 2.8 (2.84)
  Visit 17/Day 71: number analyzed (Participants) | 56 | 48
  Visit 17/Day 71 | 2.4 (2.13) | 2.3 (2.35)
  Visit 18/Day 78: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78 | 2.1 (1.97) | 1.9 (1.96)

11. Secondary Outcome: Ovarian Follicular Activity Measured by the Maximum Diameter of the Largest Ovarian Follicle
Description: Maximum diameter of largest ovarian follicle measured at Baseline, Visits 1-10, Visits 12-18 (Days 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78)
Time Frame: Days 0, 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, up to 78 days
Population: Subjects that had follicles measured and counted were analyzed
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
mm
  Baseline: number analyzed (Participants) | 55 | 54
  Baseline | 15.9 (6.00) | 16.1 (6.09)
  Visit 1/Day 1: number analyzed (Participants) | 45 | 50
  Visit 1/Day 1 | 9.9 (3.60) | 10.4 (5.27)
  Visit 3/Day 5: number analyzed (Participants) | 55 | 51
  Visit 3/Day 5 | 13.0 (4.08) | 12.9 (6.46)
  Visit 4/Day 8: number analyzed (Participants) | 54 | 53
  Visit 4/Day 8 | 16.0 (5.34) | 16.0 (7.35)
  Visit 5/Day 11: number analyzed (Participants) | 55 | 54
  Visit 5/Day 11 | 16.1 (7.13) | 17.4 (7.85)
  Visit 7/Day 18: number analyzed (Participants) | 56 | 51
  Visit 7/Day 18 | 15.1 (9.71) | 18.8 (11.76)
  Visit 8/Day 22: number analyzed (Participants) | 38 | 45
  Visit 8/Day 22 | 16.6 (11.64) | 17.3 (10.96)
  Visit 9/Day 25: number analyzed (Participants) | 43 | 46
  Visit 9/Day 25 | 15.0 (9.80) | 18.8 (12.82)
  Visit 10/Day 29: number analyzed (Participants) | 52 | 47
  Visit 10/Day 29 | 12.9 (8.51) | 17.0 (11.94)
  Visit 12/Day 36: number analyzed (Participants) | 53 | 48
  Visit 12/Day 36 | 16.0 (7.55) | 18.1 (11.34)
  Visit 13/Day 43: number analyzed (Participants) | 51 | 44
  Visit 13/Day 43 | 16.2 (9.35) | 18.5 (9.83)
  Visit 14/Day 50: number analyzed (Participants) | 43 | 46
  Visit 14/Day 50 | 16.1 (10.49) | 16.7 (8.23)
  Visit 15/Day 57: number analyzed (Participants) | 50 | 46
  Visit 15/Day 57 | 16.9 (11.06) | 14.5 (7.41)
  Visit 16/Day 64: number analyzed (Participants) | 52 | 42
  Visit 16/Day 64 | 18.3 (10.36) | 13.5 (6.80)
  Visit 17/Day 71: number analyzed (Participants) | 50 | 38
  Visit 17/Day 71 | 17.9 (11.60) | 16.5 (8.13)
  Visit 18/Day 78: number analyzed (Participants) | 47 | 40
  Visit 18/Day 78 | 16.7 (11.32) | 16.8 (9.58)

12. Secondary Outcome: Ovarian Follicular Activity Measured by the Average Diameter of the Largest Ovarian Follicle
Description: Average diameter of largest ovarian follicle measured at Baseline, Visits 1-10, Visits 12-18 (Days 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78)
Time Frame: Days 0, 1, 5, 8, 11, 18, 22, 25, 29, 36, 43, 50, 57, 64, 71, 78, up to 78 days
Population: Subjects that had follicles measured and counted were analyzed
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
mm
  Baseline: number analyzed (Participants) | 55 | 54
  Baseline | 14.2 (5.7) | 14.5 (5.30)
  Visit 1/Day 1: number analyzed (Participants) | 45 | 50
  Visit 1/Day 1 | 8.7 (3.34) | 9.0 (4.90)
  Visit 3/Day 5: number analyzed (Participants) | 55 | 51
  Visit 3/Day 5 | 11.8 (3.85) | 11.6 (5.98)
  Visit 4/Day 8: number analyzed (Participants) | 54 | 53
  Visit 4/Day 8 | 14.4 (5.00) | 14.5 (6.54)
  Visit 5/Day 11: number analyzed (Participants) | 55 | 54
  Visit 5/Day 11 | 14.4 (6.21) | 15.4 (7.29)
  Visit 7/Day 18: number analyzed (Participants) | 56 | 51
  Visit 7/Day 18 | 13.7 (9.08) | 16.9 (10.68)
  Visit 8/Day 22: number analyzed (Participants) | 38 | 45
  Visit 8/Day 22 | 14.4 (9.82) | 15.6 (10.14)
  Visit 9/Day 25: number analyzed (Participants) | 43 | 46
  Visit 9/Day 25 | 12.8 (8.29) | 16.8 (11.92)
  Visit 10/Day 29: number analyzed (Participants) | 52 | 47
  Visit 10/Day 29 | 11.5 (7.57) | 15.4 (10.69)
  Visit 12/Day 36: number analyzed (Participants) | 53 | 48
  Visit 12/Day 36 | 14.4 (6.88) | 16.2 (9.99)
  Visit 13/Day 43: number analyzed (Participants) | 51 | 44
  Visit 13/Day 43 | 14.3 (8.83) | 16.8 (9.04)
  Visit 14/Day 50: number analyzed (Participants) | 43 | 46
  Visit 14/Day 50 | 14.5 (9.45) | 14.8 (7.56)
  Visit 15/Day 57: number analyzed (Participants) | 50 | 46
  Visit 15/Day 57 | 14.8 (9.87) | 13.1 (6.89)
  Visit 16/Day 64: number analyzed (Participants) | 52 | 42
  Visit 16/Day 64 | 16.6 (9.70) | 11.8 (5.88)
  Visit 17/Day 71: number analyzed (Participants) | 50 | 38
  Visit 17/Day 71 | 15.7 (10.55) | 14.9 (7.45)
  Visit 18/Day 78: number analyzed (Participants) | 47 | 40
  Visit 18/Day 78 | 14.7 (10.24) | 15.1 (8.73)

13. Secondary Outcome: Number of Subjects That Possibly Ovulated (Serum Progesterone 3-10 ng/mL)
Description: Number of subjects that possibly ovulated based on serum progesterone > 3.0 ng/mL but <10 ng/mL measured during Weeks 1-4, 5-8, 9-11, and Post-Treatment Week 12
Time Frame: Weeks 1-4, 5-8, 9-11, and Post-Treatment Week 12, up to 12 weeks
Population: Subjects that had serum progesterone measured during the respective weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
Participants
  Weeks 1-4 | 14 | 15
  Weeks 5-8: number analyzed (Participants) | 59 | 56
  Weeks 5-8 | 27 | 8
  Weeks 9-11: number analyzed (Participants) | 57 | 49
  Weeks 9-11 | 16 | 7
  Post-Treatment Week 12: number analyzed (Participants) | 57 | 49
  Post-Treatment Week 12 | 18 | 10

14. Secondary Outcome: Number of Subjects That Likely Ovulated (Serum Progesterone > 10 ng/mL)
Description: Number of subjects that possibly ovulated based on serum progesterone > 10 ng/mL measured during Weeks 1-4, 5-8, 9-11, and Post-Treatment Week 12
Time Frame: Weeks 1-4, 5-8, 9-11, and Post-Treatment Week 12, up to 12 weeks
Population: Subjects that had serum progesterone measured during the respective weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 60 | 57
Participants
  Weeks 1-4 | 29 | 9
  Weeks 5-8: number analyzed (Participants) | 59 | 56
  Weeks 5-8 | 12 | 4
  Weeks 9-11: number analyzed (Participants) | 57 | 49
  Weeks 9-11 | 12 | 6
  Post-Treatment Week 12: number analyzed (Participants) | 57 | 49
  Post-Treatment Week 12 | 7 | 5

15. Secondary Outcome: Bleeding Patterns Based on Number of Bleeding/Spotting Days
Description: Bleeding and spotting days are recorded via subject diary and the number of days of bleeding and spotting are assessed during Weeks 1-4, Weeks 5-8, Weeks 5-9, and Post-Treatment Week 12
Time Frame: Weeks 1-4, Weeks 5-8, Weeks 5-9, and Post-Treatment Week 12, up to 12 Weeks
Population: subjects that completed diaries during the specified timeframe
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 61 | 60
Number of Days
  Weeks 1-4: number analyzed (Participants) | 59 | 56
  Weeks 1-4 | 7.5 (3.47) | 7.4 (3.73)
  Weeks 5-8: number analyzed (Participants) | 57 | 50
  Weeks 5-8 | 6.6 (4.53) | 9.4 (5.68)
  Weeks 9-11: number analyzed (Participants) | 57 | 49
  Weeks 9-11 | 5.1 (4.09) | 6.3 (4.71)
  Post-Treatment Week 12: number analyzed (Participants) | 12 | 19
  Post-Treatment Week 12 | 2.9 (4.27) | 2.1 (2.30)

16. Secondary Outcome: Patch Wearability Based on Skin Irritation
Description: Patch wearability measured by patch site skin irritation at Visit 4, Visit 6, Visit 8, Visit 10, Visits 12-18 (Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78) based on the following criteria: None= No irritation or barely perceptible/spotty erythema; Mild= Mild erythema covering approximately <50% of the application site; Moderate = Moderate erythema covering approximately >=50% of the application site, possible presence of mild edema; Significant = Severe erythema, possible edema, vesiculation, bullae and/or ulceration.
Time Frame: Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, up to 78 days
Population: subjects that had patch site skin irritation assessed during the respective timepoints are included
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
Number analyzed (Participants) | 61 | 60
Participants
  Visit 4/Day 8: None: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: None | 55 | 47
  Visit 4/Day 8: Mild: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: Mild | 5 | 9
  Visit 4/Day 8: Moderate: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: Moderate | 0 | 2
  Visit 4/Day 8: Significant: number analyzed (Participants) | 60 | 58
  Visit 4/Day 8: Significant | 0 | 0
  Visit 6/Day 15: None: number analyzed (Participants) | 58 | 56
  Visit 6/Day 15: None | 50 | 42
  Visit 6/Day 15: Mild: number analyzed (Participants) | 58 | 56
  Visit 6/Day 15: Mild | 7 | 13
  Visit 6/Day 15: Moderate: number analyzed (Participants) | 58 | 56
  Visit 6/Day 15: Moderate | 1 | 1
  Visit 6/Day 15: Significant: number analyzed (Participants) | 58 | 56
  Visit 6/Day 15: Significant | 0 | 0
  Visit 8/Day 22: None: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: None | 53 | 45
  Visit 8/Day 22: Mild: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: Mild | 6 | 7
  Visit 8/Day 22: Moderate: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: Moderate | 0 | 3
  Visit 8/Day 22: Significant: number analyzed (Participants) | 59 | 55
  Visit 8/Day 22: Significant | 0 | 0
  Visit 10/Day 29: None: number analyzed (Participants) | 58 | 54
  Visit 10/Day 29: None | 52 | 42
  Visit 10/Day 29: Mild: number analyzed (Participants) | 58 | 54
  Visit 10/Day 29: Mild | 5 | 9
  Visit 10/Day 29: Moderate: number analyzed (Participants) | 58 | 54
  Visit 10/Day 29: Moderate | 1 | 3
  Visit 10/Day 29: Significant: number analyzed (Participants) | 58 | 54
  Visit 10/Day 29: Significant | 0 | 0
  Visit 12/Day 36: None: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: None | 53 | 38
  Visit 12/Day 36: Mild: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: Mild | 5 | 15
  Visit 12/Day 36: Moderate: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: Moderate | 1 | 1
  Visit 12/Day 36: Significant: number analyzed (Participants) | 59 | 54
  Visit 12/Day 36: Significant | 0 | 0
  Visit 13/Day 43: None: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: None | 48 | 37
  Visit 13/Day 43: Mild: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: Mild | 8 | 14
  Visit 13/Day 43: Moderate: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: Moderate | 1 | 1
  Visit 13/Day 43: Significant: number analyzed (Participants) | 57 | 52
  Visit 13/Day 43: Significant | 0 | 0
  Visit 14/Day 50: None: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: None | 53 | 39
  Visit 14/Day 50: Mild: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: Mild | 2 | 10
  Visit 14/Day 50: Moderate: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: Moderate | 2 | 1
  Visit 14/Day 50: Significant: number analyzed (Participants) | 57 | 50
  Visit 14/Day 50: Significant | 0 | 0
  Visit 15/Day 57: None: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: None | 50 | 36
  Visit 15/Day 57: Mild: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: Mild | 6 | 10
  Visit 15/Day 57: Moderate: number analyzed (Participants) | 57 | 49
  Visit 15/Day 57: Moderate | 1 | 3
  Visit 15/Day 57: Significant: number analyzed (Participants) | 57 | 60
  Visit 15/Day 57: Significant | 0 | 0
  Visit 16/Day 64: None: number analyzed (Participants) | 56 | 49
  Visit 16/Day 64: None | 45 | 39
  Visit 16/Day 64: Mild: number analyzed (Participants) | 56 | 49
  Visit 16/Day 64: Mild | 11 | 8
  Visit 16/Day 64: Moderate: number analyzed (Participants) | 56 | 49
  Visit 16/Day 64: Moderate | 0 | 2
  Visit 16/Day 64: Significant: number analyzed (Participants) | 56 | 49
  Visit 16/Day 64: Significant | 0 | 0
  Visit 17/Day 71: None: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: None | 51 | 39
  Visit 17/Day 71: Mild: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: Mild | 4 | 6
  Visit 17/Day 71: Moderate: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: Moderate | 2 | 3
  Visit 17/Day 71: Significant: number analyzed (Participants) | 57 | 49
  Visit 17/Day 71: Significant | 0 | 1
  Visit 18/Day 78: None: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: None | 53 | 40
  Visit 18/Day 78: Mild: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: Mild | 3 | 6
  Visit 18/Day 78: Moderate: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: Moderate | 0 | 1
  Visit 18/Day 78: Significant: number analyzed (Participants) | 56 | 48
  Visit 18/Day 78: Significant | 0 | 1

ADVERSE EVENTS:
Arm/Group | Dose Level AG1000-6.5 | Dose Level AG1000-12.5
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/60
Other Adverse Events (participants affected / at risk) | 53/61 | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level AG1000-6.5 (N=61) | Dose Level AG1000-12.5 (N=60)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level AG1000-6.5 (N=61) | Dose Level AG1000-12.5 (N=60)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 5 | 5
Application site discolouration (General disorders) | 1 | 3
Application site irritation (General disorders) | 12 | 21
Fatigue (General disorders) | 1 | 3
Pain (General disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 8
Urinary tract infection (Infections and infestations) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Headache (Nervous system disorders) | 19 | 24
Breast tenderness (Reproductive system and breast disorders) | 6 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 4
Menstruation irregular (Reproductive system and breast disorders) | 5 | 7
Vaginal haemorrhage (Reproductive system and breast disorders) | 7 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 16 | 20
Acne (Skin and subcutaneous tissue disorders) | 5 | 1
Hot flush (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less